CLINICAL TRIAL: NCT00736203
Title: Memory and Picture Viewing Study
Acronym: MPVS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00008250
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-01

CONDITIONS: Healthy; Brain Reactivity of Non-smokers Undergoing fMRI Scanning
Keywords: fMRI; non-smokers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: non-smokers

SUMMARY:
The purpose of this study is to obtain a database of brain function from a sample of non-smokers while they do tasks in an MRI (magnetic resonance imaging) machine. Our hypothesis is that among nonsmokers, reactivity to smoking cues will be highly similar to control cues but may vary as a function of attitudes toward smoking and/or family history of smoking. We also hypothesize that brain activity during the n-back task will be more similar to data collected during this task when smokers are not abstinent.

DETAILED DESCRIPTION:
Thirty six non-smokers will undergo functional magnetic resonance imaging (fMRI) scanning. During scanning participants will complete the n-back task-a measure of working memory-and the cue-reactivity task-a measure of responses to smoking cues. Before scanning, participants will complete a training session where they will be familiarized with the tasks.

All participants will have to pass a screening visit in order to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* right-handed non-smokers
* between the ages of 18-55
* an expired CO concentration of 5 ppm or less; or a negative urine cotinine test of 100 ng/mL or less (to confirm a non-smoker)
* having smoked < 50 cigarettes in their lifetime

Exclusion Criteria:

* inability to attend all sessions
* significant health problems (hypertension, emphysema, seizure disorder, history of significant heart problems)
* use of psychoactive medications
* use of any tobacco or nicotine containing products
* current alcohol or drug abuse
* use of illegal drugs as measure by a urine drug screen
* presence of conditions that would make MRI unsafe (pacemaker, metallic implants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: generally healthy, right-handed non-smokers, between the ages of 18-55, having smoked less than 50 cigarettes in their lifetime
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
brain reactivity | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McClernon, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States